CLINICAL TRIAL: NCT06272188
Title: The Effect of Online Preconception Counseling on Information and Care Practices for Couples Planning Pregnancy for Healthy Beginnings
Brief Title: Preconception Care for Couples Planning Pregnancy
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Yuzuncu Yil University (Other)
Collaborators: Marmara University (Other); Kocaeli University (Other); Kastamonu University (Other); Maltepe University (Other); Izmir Katip Celebi University (Other)
Responsible Party: Principal Investigator, Esra SARI, Asist Prof., Yuzuncu Yil University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Prevention
Other Study IDs: 09.2023.1435
Record Dates: First submitted 2024-01-10; First posted 2024-02-22 (Actual); Last update posted 2024-02-22 (Actual); Status verified 2024-02

CONDITIONS: Preconception Care, Preconception Risk
Keywords: Preconceptional care; Preconceptional risk factors; Online counseling; Nursing

STUDY DESIGN:
Intervention Model Description: We do not use a model
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimantal group (Experimental): Couples applying to municipal marriage offices will be invited to participate in a study after obtaining permission. Those agreeing will be briefed by researchers about the study's purpose and methods, signing the IVCF afterward. Using a random number table, couples will be grouped as experimental or control. A month post-wedding, couples receive a call to confirm an online interview appointment. On the set date, a Zoom link for the interview will be shared. During this session, couples complete forms like IIF, PRRA, PCHLS, and PPHBS, followed by online preconception counseling lasting approximately an hour. This counseling, based on relevant literature and standardized by the research team, addresses risks identified during the Preconceptional Period Risk Assessment Form. After three months, couples revisit the PCHLS and PPHBS assessments.
  Interventions: Other: web-based online preconceptional counselling
- Control group (No Intervention): No application will be made to the control group. Note: To act ethically, online preconception care counselling will be given to the participants in the control group after the data are obtained from the experimental and control groups. In addition, the website sagliklibaslangiclar.com will be introduced and it will be explained that they will be able to log in to the website with the username and password they will be given.

INTERVENTIONS:
Other: web-based online preconceptional counselling — web-based online preconceptional counselling
  Arms: Experimantal group

SUMMARY:
Preconception care is to optimize health, address modifiable risk factors, and eliminate or reduce health-threatening factors for the woman, fetus, and newborn by working with couples to achieve a healthy pregnancy. Preconception care is the best way to protect against risks in pregnancy and plan risk management. Preconception care offers women and their partners the opportunity to gain healthy lifestyle behaviors, make conscious choices, and gain awareness of factors that threaten health before, during and after pregnancy. However, the rate of receiving preconception care is only 12.3% in our country.

The aim of this project is to examine the effect of online preconception counseling on information and care practices for couples planning pregnancy for healthy starts.

Materials and Methods:

The randomized controlled experimental study will be conducted between February 1, 2024 and February 1, 2026 in the provinces of Istanbul, Izmir, Kastamonu, Ankara and Van. The population of the research will consist of all couples who applied to the marriage offices in the above provinces between February 1, 2024 and February 1, 2026. In the sample calculation, it was calculated that at least 80 couples (experimental group: 40 couples, control group: 40 couples) should be included in the study. Couples that meet the sampling criteria will be assigned to the experimental or control group according to the random numbers table. Online preconception care counseling will be provided to couples in the experimental group 1 month after their wedding date. Preconception care counseling, consisting of 17 titles, was prepared in line with the relevant literature and standardized by the researchers. After the counseling, the couples will be introduced to the preconception care website, which they can use if they need it, and will be given login information.

Data will be obtained before and in the 3rd month after counseling with the Introductory Information Form (TBF), Preconceptional Period Risk Assessment Form, Preconceptional Care Health Literacy Scale and Preconceptional Period Health Behavior Scale. The data will be transferred to the SPSS 22 program and evaluated by the researchers. Chi-square test, t-test, Mann Whitney-U Test, Wilcoxon test and paired simple t test will be used to analyze the data.

DETAILED DESCRIPTION:
The subject of the study is preconceptional care counseling. Preconception care is a health care offered for the early detection and prevention of factors that may cause morbidity and mortality in the mother and baby during pregnancy, birth, and postnatal period. A healthy pregnancy and birth need to determine the risks by interviewing couples in the planning stage of pregnancy, to plan/implement interventions to reduce risks and to provide healthy life behaviors to couples. Preconceptional care counseling is a subject that has become increasingly important in recent years. The project is based on this issue.

Organizations such as WHO, CDC, and ACOG have reported that all couples in the preconception period should be evaluated by health professionals, and women who smoke/drink alcohol, have chronic diseases (diabetes, hypertension, hypothyroidism, epilepsy, etc.), are infected with Rubella and Hepatitis-B, have genetic diseases, have folic acid and nutritional deficiencies, are overweight and obese should be considered in the risk group in terms of maternal and fetal morbidity and mortality. It has been reported that it is essential for the protection of maternal and fetal health that all women, especially women in the risk group, receive PCC. For example, the incidence of neural tube defects such as sipina bifida and anencephaly decreases in the babies of women who start taking folic acid at least 1 month before pregnancy. Similarly, maintaining the woman's blood glucose level at normal levels during the PC period has been reported to reduce maternal morbidity, spontaneous abortion, fetal malformations, fetal macrosomia, and neonatal morbidity. Other PCC practices that protect maternal and fetal health include healthy nutrition, physical exercise, weight control, alcohol, and smoking cessation, diagnosis and treatment of chronic diseases, detection of genetic diseases, prevention of exposure to occupational and environmental agents, prevention of over-the-counter drug use, immunization, screening and prevention of infectious diseases, breast examination, dental examination, and cervical evaluation.

In recent years, there have been significant developments in the provision of preconceptional care. One of these is online preconception counseling, which is proposed to be used in this project.

Today, with the advancement of technology and the increasing importance given to education, it has become inevitable to utilize technological opportunities in solving educational problems. Written, audio, and video communication and interaction can be provided over the Internet. The education provided by using internet facilities is called "online education". Functionally, distance education provides the opportunity to learn at any time, place, amount, and speed for those who are working, busy, and want to learn what they need immediately and as much as necessary. Although there are countries in the world that have been providing online education for many years, this technology has only recently started to be used in Turkey. Internet-based education is independent of time and space, can respond to fast or slow learning needs, provides fast access to expert information and the opportunity to work with experts, provides learning opportunities that appeal to multiple senses with multimedia opportunities and reduces the cost of education. The disadvantages of online education are that the internet and computers are required, transportation is difficult in rural areas, and it may prevent socialization.

Online education is most often used in health education. Online preconception counselling is important in raising awareness of couples and helping them to develop positive health behaviors. It makes a difference in couples' understanding of their current situation. For example, in Yenal's study, the effect of web-based counseling on the activities of daily living of pregnant women was examined and 7-week training was given to pregnant women over the internet. In the study, the daily living activities scores of pregnant women gradually increased. In the study, it was found that the pregnant women continued to use the information after the end of the training.

Within the scope of the project;

1. The relevant literature was examined and it was decided to prepare and implement an online preconception care counseling program consisting of 17 topics in line with the relevant literature.
2. A website will be prepared in which information material, video, pictures, and question and answer forms will be added in parallel with the information given in online counseling.
3. To objectively evaluate the effectiveness of the online training, the "Preconceptional Period Risk Assessment Form" planned to be used in the project was prepared by the researchers, and the Turkish validity and reliability of the "Preconceptional Care Health Literacy Scale" was carried out.
4. The researchers interviewed the marriage offices where the study was planned to be carried out and obtained verbal consent. The permission letters of the institutions have been written and the response is awaited.

ELIGIBILITY:
Inclusion Criteria:

* Repuclic of Turkiye to be a citizen
* Being at least a primary school graduate
* Being over 18 years of age
* Having applied to the marriage office to get a wedding date.
* No communication barrier (such as deafness)
* Being married for the first time (both men and women having their first marriage)
* Not having experienced pregnancy
* The couple wants to have children in the future

Exclusion Criteria:

* Being under 18 years of age
* Miscarriage, abortion, stillbirth, birth, etc. Having had a pregnancy that resulted in
* Having received training on preconception care.
* Presence of a diagnosed psychiatric disease (schizophrenia, manic depressive disorder, etc.)
* Not having the necessary technological infrastructure for online consultancy.
* The woman is in menopause
* Being pregnant
* Being a healthcare worker (Doctor, Nurse, Midwife)

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 160 (Estimated)
Dates: Start 2024-02-15 (Estimated); Primary Completion 2025-07-15 (Estimated); Study Completion 2025-08-15 (Estimated)

PRIMARY OUTCOMES:
Identifying Information Form | baseline (pre intervention)
  Participants will receive web-based online preconceptional counseling.

SECONDARY OUTCOMES:
Preconceptional Period Risk Assessment Form | baseline (pre intervention)
  The preconceptional period risk assessment form, team in line with the current literature, consists of a total of 45 closed-ended questions. The form, which was finalised as a result of expert evaluations, is in the process of publication

OTHER OUTCOMES:
Preconceptional Care Health Literacy Scale | Data will be collected before preconception counselling (intervention) and three months after preconception counselling. Data will be reported no later than September 1, 2025.
  Consists of a total of 45 closed-ended questions. The form, which was finalised as a result of expert evaluations, is in the process of publication.
Preconceptional Period Health Behavior Scale | The preconceptional Period Health Behavior Scale will be used to collect data during the pre-intervention phase and the third month after the intervention.
  PDSS, which evaluates health behaviors in the preconception period, has a total of 18 items. Turan et al. (2022) consists of four sub-dimensions. Sub-dimensions are 'Preparation' (items 1,2,3,4,5,6,7 and 8), 'Coping Skills' (items 9,10 and 11), 'Risky Behaviors' (items 12,13 and 14th item) and 'Nutrition and Sleep' 15,16,17 and 18th items) sub-dimensions.
  The PDSS score is calculated by summing the scores in the answers to 18 statements. Item answers are 'Yes', 'Partly' and 'No'. "2" points are given for "Yes", "1" point is given for "Partly" and "0" points are given for "No". Accordingly, the highest total score obtained from the scale is 36, and the lowest score is 'zero'. The minimum and maximum scores for the sub-dimensions are as follows; It is 0-16, 0-6, 0-6 and 0-8 points. High scale and subscale scores indicate that women's preconception period health behaviors are positive.

CONTACTS AND LOCATIONS:
Overall Officials: Ozlem Can Gurkan, Study Director — Marmara University; Eda Simsek Sahin, Principal Investigator — Kocaeli University
Locations (1):
- Van Yuzuncu Yil University, Van, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No